CLINICAL TRIAL: NCT04292509
Title: Risk for Ketonaemia in Type 1 Diabetes Pregnancies With Sensor-augmented Pump Therapy With Predictive Stop Before Low Compared to Stop on Low: an Open-label Crossover RCT
Brief Title: Risk for Ketonaemia in Type 1 Diabetes Pregnancies With Sensor-augmented Pump Therapy
Acronym: ROKSANA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ROKSANA study
Record Dates: First submitted 2020-02-25; First posted 2020-03-03 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Pregnant Women With Type 1 Diabetes

STUDY DESIGN:
Intervention Model Description: open-label cross-over RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAP with predictive stop before low (Experimental): Sensor-augmented pump therapy with the use of the predictive stop before low mode of action
  Interventions: Device: SAP with stop before low
- SAP with stop on low (Active Comparator): Sensor-augmented pump therapy with the use of the predictive stop on low mode of action
  Interventions: Device: SAP with stop on low

INTERVENTIONS:
Device: SAP with stop before low — cross-over comparison from stop on low to stop before low
  Arms: SAP with predictive stop before low
Device: SAP with stop on low — cross-over comparison from stop before low to stop on low
  Arms: SAP with stop on low

SUMMARY:
The ROKSANA study is an open-label crossover RCT with the aim to evaluate whether sensor-augmented pump therapy (SAP) with predictive low glucose suspend technology is associated with an increased risk for ketonaemia during type 1 diabetes pregnancies.

DETAILED DESCRIPTION:
10 pregnant women with type 1 diabetes will be included . Participants will be randomized 1/1 between 12-30 weeks of pregnancy to SAP with predictive stop before low during two weeks or predictive stop on low. Participants will be cross-over to the other group after two weeks (from stop before low to stop on low or vice versa). During the study, participants will be asked to measure blood ketones three times per day.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes
* age 18-45 years
* a singleton pregnancy with ultrasound-confirmed gestational age between 12- 30 weeks.
* treated with 640 insulin pump and have a baseline HbA1c level ≤10%.

Exclusion Criteria:

* a physical or psychological disease likely to interfere with the conduct of the study
* medications known to interfere with glucose metabolism

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
blood ketones > 0.6mmol/l. | 4 weeks
  ketonaemia

SECONDARY OUTCOMES:
mean concentration of blood ketones | 4 weeks
mean time of suspension of insulin delivery | 4 weeks
frequency of hospitalization due to ketonaemia | 4 weeks
mean glucose based on CGM | 4 weeks
time >140 mg/dl | 4 weeks
time >180 mg/dl | 4 weeks
time <63 mg/dl | 4 weeks
time <50mg/dl | 4 weeks
coefficient of variation of glycaemic measurements | 4 weeks
standard deviation of glycaemic measurements | 4 weeks
mean amplitude of glucose excursions | 4 weeks
HbA1c | 4 weeks
time 70-180 mg/dL | 4 weeks
frequency of CGM use >80% of time | 4 weeks
  CGM compliance
total insulin dose | 4 weeks
severe hypoglycemic episodes | 4 weeks
  defined as requiring third-party assistance and/or capillary glucose <50 mg/dL associated with clinical symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Katrien Benhalima, MD PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benhalima K, van Nes F, Laenen A, Gillard P, Mathieu C. Risk for ketonaemia in type 1 diabetes pregnancies with sensor-augmented pump therapy with predictive low glucose suspend compared with low glucose suspend: a crossover RCT. Diabetologia. 2021 Dec;64(12):2725-2730. doi: 10.1007/s00125-021-05589-y. Epub 2021 Oct 13. PMID 34647140